CLINICAL TRIAL: NCT01382095
Title: A Phase 1 Dose-Escalating Study of dscCfaE, Co-Administered With and Without LTR192G, by Transcutaneous Immunization (TCI) in Healthy Adult U.S. Volunteers
Brief Title: Safety Study of Recombinant Vaccine to Prevent ETEC Diarrhea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A-16682; NMRC.2011.0004 (Other: Naval Medical Research Center); WRAIR 1804 (Other: Walter Reed Army Institute of Research)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Escherichia Coli Infection
Keywords: ETEC; Diarrhea; Vaccine
MeSH Terms: conditions — Escherichia coli Infections; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental)
  Interventions: Biological: Recombinant fimbrial adhesin dscCfaE; Biological: Modified E. coli heat labile enterotoxin LTR192G
- Group B-1 (Experimental)
  Interventions: Biological: Recombinant fimbrial adhesin dscCfaE; Biological: Modified E. coli heat labile enterotoxin LTR192G
- Group B-2 (Experimental)
  Interventions: Biological: Recombinant fimbrial adhesin dscCfaE
- Group C (Experimental)
  Interventions: Biological: Recombinant fimbrial adhesin dscCfaE; Biological: Modified E. coli heat labile enterotoxin LTR192G

INTERVENTIONS:
Biological: Recombinant fimbrial adhesin dscCfaE — 10 ug on study days 0, 21 and 42
  Other Names: dscCfaE
  Arms: Group A
Biological: Recombinant fimbrial adhesin dscCfaE — 50 ug on study days 0, 21 and 42
  Other Names: dscCfaE
  Arms: Group B-1; Group B-2
Biological: Recombinant fimbrial adhesin dscCfaE — 250 ug on study days 0, 21 and 42
  Other Names: dscCfaE
  Arms: Group C
Biological: Modified E. coli heat labile enterotoxin LTR192G — 50 ug on study days 0, 21 and 42
  Other Names: LTR192G
  Arms: Group A; Group B-1; Group C

SUMMARY:
The purpose of the study is to determine if immunization with a recombinant E. coli protein, dscCfaE, is safe and immunogenic when administered through the skin using a patch.

DETAILED DESCRIPTION:
The purpose of the study is to determine if immunization with dscCfaE with or without a modified E. coli heat labile enterotoxin, LTR192G, is safe and immunogenic when administered transcutaneously using a skin wet-patch. If the vaccine is found safe and adequately immunogenic in humans, a phase 2b vaccination/challenge study would be undertaken to further evaluate vaccine safety and allow a preliminary assessment of efficacy. With favorable evidence for safety, immunogenicity, efficacy, complemented by advances in standard methodology to combine multiple adhesins with an appropriate LT enterotoxoid form, a multivalent vaccine would be constructed and evaluated for further clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, age 18 to 45 years (inclusive) at the time of enrollment.
* Completion and review of comprehension test (achieved > 70% accuracy).
* Signed informed consent document.
* Available for the required follow-up period and scheduled clinic visits.
* Women: Negative pregnancy test with understanding (through informed consent process) to not become pregnant during the study or within three (3) months following study completion.

Exclusion Criteria:

* Health problems such as, chronic medical conditions such as psychiatric conditions, diabetes mellitus, hypertension or any other conditions that might place the volunteer at increased risk of adverse events. Study clinicians, in consultation with the principal investigator (PI), will use clinical judgment on a case-by-case basis to assess safety risks under this criterion. The PI will consult with the Medical Monitor as appropriate.
* Clinically significant abnormalities on physical examination.
* Immunosuppressive drugs (use of systemic corticosteroids or chemotherapeutics that may influence antibody development) or illness (including IgA deficiency).
* Women who are pregnant or planning to become pregnant during the study period plus 3 months beyond the last study safety visit and currently nursing women.
* Participation in research involving another investigational product (defined as receipt of investigational product or exposure to invasive investigational device) 30 days before planned date of first vaccination or anytime through the last study safety visit.
* Positive blood test for HBsAg, HCV, HIV-1.
* Clinically significant abnormalities on basic laboratory screening.
* Immunosuppressive illness or IgA deficiency (below the normal limits).
* Exclusionary skin history/findings that would confound assessment or prevent appropriate local monitoring of adverse events (AEs), or possibly increase the risk of an AE.
* History of chronic skin disease (clinician judgment).
* History of atopy.
* Acute skin infection/eruptions on the upper arms including fungal infections, severe acne or active contact dermatitis.
* Allergies that may increase the risk of AEs.
* Regular use (weekly or more often) of antidiarrheal, anti-constipation, or antacid therapy.
* Abnormal stool pattern (fewer than 3 stools per week or more than 3 stools per day) on a regular basis; loose or liquid stools on other than an occasional basis.
* History of microbiologically confirmed Enterotoxigenic E. coli (ETEC) or V. cholerae infection.
* Travel to countries where ETEC or V. cholerae or other enteric infections are endemic (most of the developing world) within two years prior to dosing (clinician judgment).
* Received previous experimental ETEC or V. cholerae vaccine or live ETEC or V. cholerae challenge.
* Occupation involving handling of ETEC or V. cholerae currently, or in the past 3 years.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Days 0 - 180
  Adverse event monitoring will survey and specifically inquire about fever (oral temperature > 100.4 o F), malaise, headache, rash, pain, diarrhea, abdominal pain, extremity pain or swelling. Clinical definitions will be used to grade severity of symptoms in accordance to the severity scale below: Grade 0 = None Grade 1= Barely noticeable Grade 2= Noticeable, does not interfere with daily activities Grade 3=Interferes with daily activities Grade 4=Prevents daily activities

SECONDARY OUTCOMES:
Number of Seroconversion to LT and dscCfaE; defined as a > 4-fold increase in endpoint titer between pre-and post-vaccination samples. | Study Days 0 - 180
Number of Mucosal responses (fecal IgA); defined as a > 4-fold increase in endpoint titer after adjusting for total IgA. | Study Days 0 - 180
Number of positive IgA-ASC responses; defined as a > 2-fold increase over th e baseline value of the ASC per 10 6 PBMC, when the number of ASC is > 0.5 per 10 6 in the baseline sample | Study Days 0 - 180
  A positive IgA-ASC response will be defined as a > 2-fold increase over th e baseline value of the ASC per 10 6 PBMC, when the number of ASC is > 0.5 per 10 6 in the baseline sample. When the number of baseline ASCs is less than 0.5 per 10 6 PBMC, a subject will be considered a responder if the post-vaccination value is greater than 1.0 per 10 6 PBMC

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Riddle, MD, DrPH, Principal Investigator — Naval Medical Research Center
Locations (1):
- Walter Reed Army Institute of Research Clinical Trial Center, Silver Spring, Maryland, United States